CLINICAL TRIAL: NCT00149409
Title: Omega-3-Polyunsaturated Fatty-Acids (N3-Pufa) In Patients With Severe Chronic Heart Failure:Effects On Endothelial Function, Left Ventricular Remodelling, Natriuretic Peptide Levels, And Exercise Capacity
Brief Title: Omega-3-Polyunsaturated Fatty-Acids (N3-Pufa) In Patients With Severe Chronic Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: n3-PUFA-HF
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): 4 gelatine capsules/d
  Interventions: Dietary Supplement: Omacor
- 1g/d Omacor (Active Comparator)
  Interventions: Dietary Supplement: Omacor
- 4g/d Omacor (Active Comparator)
  Interventions: Dietary Supplement: Omacor

INTERVENTIONS:
Dietary Supplement: Omacor

SUMMARY:
To investigate whether n3-fatty acids have beneficial effects in chronic heart failure as regards circulatory function.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure of non-ischemic origin
* Age ≥18 years
* NYHA functional class III-IV
* LVEF < 35 %
* Optimized heart failure therapy
* plasma NT-BNP >2000pg/ml

Exclusion Criteria:

* Current treatment with Omacor or other fish oil products
* Known hypersensitivity to the study drug
* Ischemic cardiomyopathy
* Uncorrected significant valvular heart disease
* Heart failure due to congenital heart disease
* Restrictive cardiomyopathy
* Alcoholic heart disease
* Acute myocarditis
* Continuous i.v. therapy for heart failure
* Mechanical assist device
* Life expectancy <1 year due to non-cardiac causes
* Inability to perform bicycle testing
* Women of childbearing potential not practicing a save contraception method
* Current participation in another intervention study
* Participation in another study with an intervention within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Berger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Moertl D, Hammer A, Steiner S, Hutuleac R, Vonbank K, Berger R. Dose-dependent effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of nonischemic origin: a double-blind, placebo-controlled, 3-arm study. Am Heart J. 2011 May;161(5):915.e1-9. doi: 10.1016/j.ahj.2011.02.011. PMID 21570522